CLINICAL TRIAL: NCT00525187
Title: Onychomycosis: Diagnosis and Prevalence in Diabetic Neuropathic Patients
Status: Completed | Type: Observational
Sponsor: Vésale Hospital (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Other Study IDs: Onychomycosis
Record Dates: First submitted 2007-08-20; First posted 2007-09-05 (Estimated); Last update posted 2007-09-05 (Estimated); Status verified 2007-08

CONDITIONS: Prevalence of Onychomycosis; Diabetic Neuropathic Patients; Diagnostic of Onychomycosis; Patients Clinically Suspected of Onychomycosis; Reliability of the Diagnosis of Onychomycosis
Keywords: onychomycosis; diabetic neuropathic patients; reliability of the diagnostic of onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The prevalence of onychomycosis among diabetic patients is still a debated question as well as the best way to diagnose the disease. We conducted a prospective study to assess the prevalence of onychomycosis in diabetic neuropathic (DN) patients clinically suspected of this disease and to assess the reliability of the diagnosis of onychomycosis.

DETAILED DESCRIPTION:
From December 2000 to January 2005, we followed 100 successive diabetic patients, type 1 and type 2, suffering from (DN). At baseline we assessed age, gender, medical history and medications, foot insensitivity defined by a vibration perception threshold (VPT) >25 volts and onychomycosis by clinical diagnosis.

Multiple samples of the most affected nail, often the big toe, were taken. A potassium hydroxide (KOH) test was done by 2 independent and blinded investigators and a culture in a laboratory (lab) specialized in mycology.

Pictures of the nails and particularly of the sampled nail were taken. Apart from the laboratory results, two independent and blinded dermatologists gave their diagnosis looking at the pictures.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were: presence of diabetes mellitus, type 1 or type 2, age between 18 and 80 years, neuropathy demonstrated by a VPT (Vibration Perception Threshold) >25 volts tested with a neurothesiometer (Horwell Scientific, London, UK) and a clinical diagnosis of onychomycosis.

Exclusion Criteria:

* Exclusion criteria were a history of psoriasis, systemic antifungal therapy during the year preceding the enrolment, immunosuppression either by disease or treatment induced.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-12; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle J DUMONT, MD, Principal Investigator
Locations (1):
- CHU A Vésale, Montigny-le-Tilleul, Hainaut, Belgium